CLINICAL TRIAL: NCT03277352
Title: A Phase 1/2 Safety and Efficacy Study of INCAGN01876 in Combination With Immune Therapies in Subjects With Advanced or Metastatic Malignancies
Brief Title: INCAGN01876 in Combination With Immune Therapies in Subjects With Advanced or Metastatic Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to emergent data from another study and unrelated to safety.
Sponsor: Incyte Biosciences International Sàrl (Industry)
Responsible Party: Sponsor
Organization: Incyte Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCAGN 1876-202
Record Dates: First submitted 2017-08-14; First posted 2017-09-11 (Actual); Results first posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-06

CONDITIONS: Advanced Malignancies; Metastatic Cancer
Keywords: cervical cancer; endometrial cancer; gastric cancer (including stomach and gastroesophageal junction (GEJ)); esophageal cancer; hepatocellular carcinoma (HCC); melanoma (mucosal or cutaneous); Merkel cell carcinoma; mesothelioma; microsatellite instability-high (MSI-H); solid tumors; non-small cell lung cancer (NSCLC); ovarian cancer; squamous cell carcinoma of the head and neck (SCCHN); small cell lung cancer (SCLC); renal cell carcinoma (RCC); triple-negative breast cancer (TNBC); urothelial carcinoma; glucocorticoid-induced tumor necrosis factor receptor (GITR)
MeSH Terms: conditions — Neoplasm Metastasis; Uterine Cervical Neoplasms; Endometrial Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Carcinoma, Hepatocellular; Melanoma; Carcinoma, Merkel Cell; Mesothelioma; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Squamous Cell Carcinoma of Head and Neck; Small Cell Lung Carcinoma; Carcinoma, Renal Cell; Triple Negative Breast Neoplasms; Carcinoma, Transitional Cell | interventions — epacadostat; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- INCAGN01876 + Pembrolizumab + Epacadostat (Experimental): INCAGN01876 in combination with pembrolizumab and epacadostat
  Interventions: Drug: INCAGN01876; Drug: Epacadostat; Drug: Pembrolizumab

INTERVENTIONS:
Drug: INCAGN01876 — In Phase 1 subjects will receive INCAGN01876 administered intravenously (IV) at the protocol-defined dose and schedule according to cohort and treatment group enrollment. In Phase 2, subjects will be administered IV study drug at the recommended dose from Phase 1.
Drug: Epacadostat — Epacadostat will be self-administered orally at the protocol-defined dose.
  Other Names: INCB024360
Drug: Pembrolizumab — Pembrolizumab will be administered IV at the protocol-defined dose.
  Other Names: Keytruda®

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and efficacy of INCAGN01876 when given in combination with immune therapies.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic disease; locally advanced disease must not be amenable to resection with curative intent.
* Phase 1: Subjects with advanced or metastatic solid tumors.
* Phase 1: Subjects who have disease progression after treatment with available therapies.
* Phase 2: Subjects with advanced or metastatic melanoma, RCC, and urothelial carcinoma.
* Presence of measurable disease based on RECIST v1.1.
* Eastern Cooperative Oncology Group performance status of 0 or 1.

Exclusion Criteria:

* Laboratory and medical history parameters not within the Protocol-defined range
* Prior treatment with any tumor necrosis factor super family agonist.
* Receipt of anticancer medications or investigational drugs within protocol-defined intervals before the first administration of study drug.
* Has not recovered to ≤ Grade 1 from toxic effects of prior therapy.
* Active autoimmune disease.
* Known active central nervous system metastases and/or carcinomatous meningitis.
* Evidence of active, noninfectious pneumonitis or history of interstitial lung disease.
* Evidence of hepatitis B virus or hepatitis C virus infection or risk of reactivation.
* Known history of human immunodeficiency virus (HIV; HIV 1/2 antibodies).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John N. Janik, MD, Study Director — Incyte Corporation
Locations (2):
- United States (2):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - Hackensack University Medical Center, Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 2 different sites in USA. A total of 10 participants were enrolled in the study.
Pre-assignment Details: A total of 10 participants were screened and enrolled in the study.
Period: Overall Study
Arm/Group | INCAGN01876 + Pembrolizumab + Epacadostat
Started | 10
Completed | 0
Not Completed | 10
Not completed — Study Terminated By Sponsor | 2
Not completed — Withdrawal by Subject | 4
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) includes all subjects enrolled in the study who received at least 1 dose of INCAGN01876, pembrolizumab, or epacadostat.
Arm/Group | INCAGN01876 + Pembrolizumab + Epacadostat
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (13.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 8
  Asian | 1
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 and Phase 2: Participants With Treatment-Emergent Adverse Events (TEAEs) [Safety and Tolerability]
Description: A TEAE is any adverse event (AE) either reported for the first time or worsening of a pre-existing event after the first dose of study treatment.
Time Frame: Screening through 60 days after end of treatment, up to approximately 18 months
Population: The FAS includes all participants enrolled in the study who received at least 1 dose of INCAGN01876, pembrolizumab, or epacadostat.
Measure: Count of Participants; unit: Participants
Arm/Group | INCAGN01876 + Pembrolizumab + Epacadostat
Number analyzed (Participants) | 10
Participants | 10

2. Primary Outcome: Phase 1 and Phase 2 : ORR Based on RECIST v1.1 and mRECIST
Description: Defined as the percentage of participants having a CR or PR based on investigator assessment per RECIST v1.1.
Time Frame: Assessed every 9 weeks for 12 months, then every 12 weeks, up to 18 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | INCAGN01876 + Pembrolizumab + Epacadostat
Number analyzed (Participants) | 10
Participants | 3

3. Primary Outcome: Phase 2: Complete Response Rate (CRR) Based on RECIST v1.1
Description: Defined as the percentage of checkpoint inhibitor-naive melanoma participants who have a CR based on investigator assessment per RECIST v1.1
Time Frame: Assessed every 9 weeks for 12 months, then every 12 weeks, up to 18 months
Population: The study was terminated early and no participants enrolled in Phase 2 of the study.
Arm/Group | INCAGN01876 + Pembrolizumab + Epacadostat
Number analyzed (Participants) | 0

4. Secondary Outcome: Phase 1 & Phase 2: Disease Control Rate Based on RECIST v1.1 and mRECIST
Description: Defined as the percentage of participants having CR, PR, or stable disease (SD) based on investigator assessment per RECIST v1.1.
Time Frame: Assessed every 9 weeks for 12 months, then every 12 weeks, up to 18 months.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | INCAGN01876 + Pembrolizumab + Epacadostat
Number analyzed (Participants) | 10
Participants | 7

5. Secondary Outcome: Phase 1 & Phase 2: Duration of Response Based on RECIST v1.1 and mRECIST
Description: Defined as the time from the earliest date of disease response (CR or PR) until earliest date of disease progression or death due to any cause.
Time Frame: Assessed every 9 weeks for 12 months, then every 12 weeks, up to 18 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | INCAGN01876 + Pembrolizumab + Epacadostat
Number analyzed (Participants) | 10
days | NA [273 to NA] — The median duration of response is not estimable if less than half of the participants had an event (progression or death).

6. Secondary Outcome: Phase 1 & Phase 2: Duration of Disease Control Based on RECIST v1.1 and mRECIST
Description: Defined as time from first report of SD or better until disease progression or death from any cause.
Time Frame: Assessed every 9 weeks for 12 months, then every 12 weeks, up to 18 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | INCAGN01876 + Pembrolizumab + Epacadostat
Number analyzed (Participants) | 10
days
  mRECIST | NA [525 to NA] — The median duration of response is not estimable if less than half of the participants had an event (progression or death).
  RECIST | 525 [92 to NA] — The number of responders is not enough to estimate a standard error for the confidence interval.

7. Secondary Outcome: Phase 1 & Phase 2: Progression-free Survival Based on RECIST v1.1 and mRECIST
Description: Defined as the time from the start of combination therapy until the earliest date of disease progression or death due to any cause.
Time Frame: Assessed every 9 weeks for 12 months, then every 12 weeks, up to 18 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | INCAGN01876 + Pembrolizumab + Epacadostat
Number analyzed (Participants) | 10
months
  mRECIST | 17.36 [2.05 to NA] — The number of responders is not enough to estimate a standard error for the confidence interval.
  RECIST | 4.20 [0.73 to NA] — The number of responders is not enough to estimate a standard error for the confidence interval.

8. Secondary Outcome: Phase 1 & Phase 2: Overall Survival
Description: Defined as the time from the start of combination therapy until death due to any cause.
Time Frame: At 1 year and 2 years.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | INCAGN01876 + Pembrolizumab + Epacadostat
Number analyzed (Participants) | 10
months | 25.59 [16.76 to NA] — upper limit is not estimable

ADVERSE EVENTS:
Time Frame: up to 18 months
Groups:
- INCAGN01876 300 mg Q3W + Pembrolizumab 200 mg Q3W + Epacadostat 100 mg BID: INCAGN01876 300 mg Q3W + Pembrolizumab 200 mg Q3W + Epacadostat 100 mg BID
- Total: Total
Arm/Group | INCAGN01876 300 mg Q3W + Pembrolizumab 200 mg Q3W + Epacadostat 100 mg BID | Total
All-Cause Mortality (participants affected / at risk) | 4/10 | 4/10
Serious Adverse Events (participants affected / at risk) | 3/10 | 3/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INCAGN01876 300 mg Q3W + Pembrolizumab 200 mg Q3W + Epacadostat 100 mg BID (N=10) | Total (N=10)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Uveitis (Eye disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INCAGN01876 300 mg Q3W + Pembrolizumab 200 mg Q3W + Epacadostat 100 mg BID (N=10) | Total (N=10)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Axillary pain (General disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Eye irritation (Eye disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 3 (4) | 3 (4)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1)
Hydrogen breath test abnormal (Investigations) | 1 (1) | 1 (1)
Hyperchloraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Lipase increased (Investigations) | 2 (2) | 2 (2)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Macular hole (Eye disorders) | 1 (1) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (4)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Rash generalised (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 2 (2) | 2 (2)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement

DOCUMENTS (2):
  • Study Protocol (2017-08-24): https://cdn.clinicaltrials.gov/large-docs/52/NCT03277352/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT03277352/SAP_001.pdf